CLINICAL TRIAL: NCT00858130
Title: Optimal Intensity and Frequency of a Portable Electrical Muscle Stimulator (VeinoPlus) to Improve Symptoms of Postthrombotic Syndrome
Brief Title: Pilot Study for VeinoPlus to Improve Symptoms of Postthrombotic Syndrome (PTS)
Acronym: VeinoPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: VeinoPlus USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-2143Veinoplus
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-08

CONDITIONS: Post Thrombotic Syndrome; Deep Vein Thrombosis; Venous Stasis Syndrome; Venous Insufficiency; Postphlebitic Syndrome
Keywords: Veinoplus; post thrombotic syndrome; deep vein thrombosis; electrical muscle stimulator; Venous stasis syndrome; venous insufficiency syndrome; Postphlebitic syndrome; history of deep vein thrombosis
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis; Venous Insufficiency; Postphlebitic Syndrome

STUDY DESIGN:
Intervention Model Description: Patients were told to use different voltages and numbers of treatment periods, and experiment with pad placement, to find intensity, frequency of use, and pad position for optimal PTS symptom relief. Assessments (Villalta score, QOL questionnaire, calf circumference) were obtained at study entry and after 8 weeks of device use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Veinoplus (Experimental): Every subject enrolled in study will be in this experimental arm. VeinoPlus device will be used by all enrolled subjects.
  Interventions: Device: VeinOPlus

INTERVENTIONS:
Device: VeinOPlus — The Veinoplus® device electrically stimulates leg muscles via motor nerves, causing calf muscle contractions. The two electrodes are placed on the central part of the calf muscle on the back of the legs, and once the device is turned on, the length of treatment is 20 minutes. The device has a variable intensity setting which allows subjects to choose their own level and change the stimulations mid-cycle if desired. Subjects will use the device however they see fit for 2 months.

SUMMARY:
The investigators plan to perform an exploratory study to investigate the effects of electro-stimulation of the legs on the symptoms and clinical findings of post thrombotic syndrome (PTS), as well as quality of life of patients with PTS. The investigators theorize that electro-stimulation will provide both a mechanical benefit via muscular contraction and increased venous outflow from the affected extremity, as well as an anesthetic effect, which the investigators anticipate will translate into improved symptomatic outcomes, quality of life (QOL) benefits.

DETAILED DESCRIPTION:
The purpose of this study is to determine the optimal electrical stimulation intensity level at which subjects using the portable electrical muscle stimulator (VeinoPlus) have the largest benefit for relief of post thrombotic symptoms. To determine if the subjects reported benefit from the device and willingness to continue using the device.

Subjects will be pre-screened on the phone for eligibility, and an initial appointment will be set. The subject will be given a device and complete a quality of life survey. The subject will also be assessed on the Villalta scale. After two months, the subjects will return for the final visit where the Villalta scale and quality of life survey will be reassessed, and the device taken back.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Presence of previously objectively documented unilateral, lower extremity deep venous thrombosis
* Presence of PTS (typical pain and swelling - worse after standing and vertical activity and relieved by rest and the horizontal position), severe enough that the patient is interested to explore a treatment option that might improve these symptoms. Symptoms had to have been stable for ≥ 3 months. Unstable symptoms are defined as: worsening, improving or variable symptoms over preceding months.
* Subjects must be willing and able to give written informed consent.

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Pregnancy
* Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
* Geographic inaccessibility to prevent scheduled return evaluations
* Incapable of responding to questionnaires
* Expected lifespan <6 months
* Presence of cardiac pacemaker
* History of cardiac arrhythmia
* Presence of infected, or inflamed areas or skin eruptions; phlebitis, thrombophlebitis, active venous ulceration
* History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Moll, MD, Principal Investigator — UNC Chapel Hill, Department of Medicine, Division of Hematology/Oncology
Locations (1):
- University of North Carolina at Chapel Hill; University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VeinoPlus
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 54 [21 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Leg Calf Circumference [Median (Full Range); unit: centimeters (cm)] — Leg measurements around the largest part of both calves were taken.
  centimeters (cm) | 41 [33 to 51]
Villalta Scale [Median (Full Range); unit: units on a scale] — The Villalta PTS scale is based on patient symptoms including cramps, pain, and redness. The severity of PTS was categorized using the Villalta scale. Points are given for 11 descriptors according to severity ranging from 0 (not present) to 3 (severe) with overall scores from 0 to 33. Higher scores represent more severe disease. A score of ≥ 5 indicated mild PTS, 10-14 moderate PTS, and a score of ≥ 15, or the presence of a venous ulcer, indicated severe PTS.
  units on a scale | 13 [6 to 22]
VEINES-Quality of Life (QOL) [Median (Full Range); unit: units on a scale] — The VEINES-QOL/Sym Questionnaire is a patient-based questionnaire designed for self-completion and measures the impact of deep venous thrombosis (DVT) on symptoms and quality of life from the patient's perspective. It contains 26 items covering symptoms, limitations in daily activities, and psychological impact of patients with a DVT. Summary scores are generated for disease specific quality of life (VEINES-QOL) and venous symptoms (VEINES-Sym) each ranging from 0 to 100. For the VEINES-QOL, higher scores indicate a better quality of life.
  units on a scale | 48.30 [31.11 to 57.46]
VEINES-Sym [Median (Full Range); unit: units on a scale] — The VEINES-QOL/Sym Questionnaire is a patient-based questionnaire designed for self-completion and measures the impact of deep venous thrombosis (DVT) on symptoms and quality of life from the patient's perspective. It contains 26 items covering symptoms, limitations in daily activities, and psychological impact of patients with a DVT. Summary scores are generated for disease specific quality of life (VEINES-QOL) and venous symptoms (VEINES-Sym) each ranging from 0 to 100. For the VEINES-Sym, higher scores indicate better outcomes.
  units on a scale | 46.93 [36.67 to 58.41]

OUTCOME MEASURES:

1. Primary Outcome: Median Optimal Electrical Stimulation Intensity Level for Largest Benefit in Relief of Symptoms
Description: The VeinoPlus® electrically stimulates leg muscles via motor nerves, causing muscle contractions. Two electrode pads are placed on the skin of the leg. Pad positions can be chosen by the patient, such as (a) both pads on the calf muscle of one leg, (b) one pad on the calf muscle and one on the plantar aspect of the foot of one leg, and (c) a pad posteriorly on each calf. Length of treatment is programmed into the device and is 20 minutes. The device has a variable intensity setting which allows subjects to choose their own level and change the stimulations during the treatment cycle if desired. The intensity ranges from zero to fifty, with zero being no electrical stimulation, and fifty the highest intensity, which carries low quantities of electrical energy (<5 micro coulombs). In this study subjects used the device at any setting, as many times a day as they liked, and varying the placement of the electrodes.
Time Frame: Visit 2 (Week 8)
Measure: Median (Full Range); unit: mirco coulombs (0 to 50)
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
mirco coulombs (0 to 50) | 32 [20 to 40]

2. Secondary Outcome: Number of Study Participants Classified as a "Clinical Success"
Description: Clinical success was defined by the patient reporting benefit (moderate improvement of symptoms after having used the device) and an interest and willingness to continue using the device. For this study both legs were measured, but only the more severely affected leg (as determined by higher Villalta score) was used to determine clinical success. Patients were asked the following question: "How much have symptoms improved?" with the following possible responses: "a little;" "moderate;" "a good deal;" "a great deal;" or "a very great deal."
Time Frame: Visit 2 (Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
Participants | 7

3. Secondary Outcome: Number of Study Participants With Improvements in PTS Severity (Villalta Score)
Description: The Villalta PTS scale is based on patient symptoms including cramps, pain, and redness and was used to characterize PTS severity. Points are given for 11 descriptors according to severity from 0 (not present) to 3 (severe) with overall scores ranging from 0 to 33. Higher scores represent more severe disease. A score of ≥ 5 indicated mild PTS; 10-14 moderate PTS; and a score of ≥15, or the presence of a venous ulcer, indicated severe PTS. Those participants with a Villalta score decrease at Visit 2 in comparison to Visit 1 were counted as having improved.
Time Frame: Visit 2 (Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
Participants | 8

4. Secondary Outcome: Number of Study Participants With Improvements in QOL (VEINES-QOL Score)
Description: The VEINES-QOL/Sym is a patient-based questionnaire designed for self-completion and measures DVT impact on symptoms and QOL from patients' perspective. It contains 26 items covering patient DVT: symptoms, limitations in daily activities, and psychological impact. Two separate summary scores are produced ranging from 0 to 100; a disease-specific QOL (VEINES-QOL) and venous symptoms (VEINES-Sym). For both the VEINES-QOL and VEINES-Sym, higher scores indicate a better QOL. Instruments were completed at Visits 1 and 2 (Follow-up). Those participants with a VEINES-QOL score increase at Visit 2 in comparison to Visit 1 were counted as having improved.
Time Frame: Vist 2 (Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
Participants | 10

5. Secondary Outcome: Number of Study Participants With Improvements in Venous Symptoms (VEINES-Sym Score)
Description: The VEINES-QOL/Sym is a patient-based questionnaire designed for self-completion and measures DVT impact on symptoms and QOL from patients' perspective. It contains 26 items covering patient DVT: symptoms, limitations in daily activities, and psychological impact. Two separate summary scores are produced ranging from 0 to 100; a disease-specific QOL (VEINES-QOL) and venous symptoms (VEINES-Sym). For both the VEINES-QOL and VEINES-Sym, higher scores indicate a better QOL. Instruments were completed at Visits 1 and 2 (Follow-up). Those participants with a VEINES-Sym score increase at Visit 2 in comparison to Visit 1 were counted as having improved.
Time Frame: Vist 2 (Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | VeinoPlus
Number analyzed (Participants) | 12
Participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire duration of study subject participation which was 8 weeks.
Groups:
- VeinoPlus Experimental Arm: Every subject enrolled in study will be in this experimental arm. VeinoPlus device will be used by all enrolled subjects.
  VeinoPlus: The VeinoPlus® device electrically stimulates leg muscles via motor nerves, causing calf muscle contractions. The two electrodes are placed on the central part of the calf muscle on the back of the legs, and once the device is turned on, the length of treatment is 20 minutes. The device has a variable intensity setting which allows subjects to choose their own level and change the stimulations mid-cycle if desired. Subjects will use the device however they see fit for 2 months.
Arm/Group | VeinoPlus Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeinoPlus Experimental Arm (N=12)
"pinhole leak" near subject's left ankle (Skin and subcutaneous tissue disorders) | 1 (1) — Subject got a "pinhole leak" near her left ankle that releases fluid. Subject has discontinued using the device on her left leg. This adverse event did not result in hospital admission or prolongation of hospitalization.

LIMITATIONS AND CAVEATS:
Given its small sample size (n=12), this study provides rationale and details needed for a larger randomized, placebo controlled, and double-blinded trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes